CLINICAL TRIAL: NCT05814211
Title: A Randomized, Open-labelled, Crossover Study Confirming Performance of a New Single-use Compact Intermittent Catheter in a Population of Adult Female Intermittent Catheter Users
Brief Title: Clinical Trial of New Intermittent Single-use Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CP348
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device - newly developed intermittent catheter (Experimental): Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (CH12 and CH14) for urinary drainage. The investigational device is for single use.
  Randomization will decide the order of investigational device/comparator device and which of the two comparator devices the subject will receive in the comparator study period.
  Interventions: Device: Investigational device - newly developed intermittent catheter
- Comparator device (#1 OR #2) (Active Comparator): SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked Coloplast products.
  Randomization will decide the order of investigational device/comparator device and which of the two comparator devices the subject will receive in the comparator study period.
  Interventions: Device: Comparator device #1 - SpeediCath Eve; Device: Comparator device #2 - SpeediCath Compact Plus Female

INTERVENTIONS:
Device: Investigational device - newly developed intermittent catheter — Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
  Arms: Investigational device - newly developed intermittent catheter
Device: Comparator device #1 - SpeediCath Eve — During comparator study period, subjects will only receive one of the comparator products. Randomization will decide which one.
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
  Arms: Comparator device (#1 OR #2)
Device: Comparator device #2 - SpeediCath Compact Plus Female — During comparator study period, subjects will only receive one of the comparator products. Randomization will decide which one.
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
  Arms: Comparator device (#1 OR #2)

SUMMARY:
A multi-centre, open-labelled, randomised, crossover design. The total study duration for the individual subject will be approximately 4 weeks, consisting of four site visits and two 2-week test periods at home. Visits 0 and 1 can be performed on the same day. For visit 2 and 3, 2 catheterisations will be performed in a hospital setting (one HCP catheterisation and one self-catheterisation) for bladder emptying and user experience assessments. Visit 1 and 2 are followed by a home-use test period, followed by visit 3 which terminates the study.

ELIGIBILITY:
Inclusion Criteria:

* Is Female
* Is at least 18 years of age and has full legal capacity
* Has signed an informed consent form
* Has used clean intermittent self-catheterisation (CISC) (CH12 or CH14) for at least one month up to inclusion
* Is using intermittent self-catheterisation for a minimum of 3 times per day for bladder emptying
* Has used a compact catheter 50% of the time (or more) for the last two weeks prior to entering the study
* Has the ability (assessed by investigator) and willingness to follow study procedures

Exclusion Criteria:

* Is participating in any other clinical study during this investigation
* Has previously participated in this study
* Has symptoms of urinary tract infection at time of inclusion, as judged by the investigator (if the patient recovers within the recruitment period, a second inclusion is allowed, under a different subject id)
* Is an individual with a history of - suspected to be - or showing signs of producing an excessive amount of mucus or large/clustered sediments or debris
* Has any known allergies towards ingredients in the investigational device
* Is pregnant
* Is breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Andersen, MD, Principal Investigator — Odense Universitetshospital
Locations (11):
- Denmark (4):
  - Rigshopsitalet, Copenhagen, København Ø
  - Sanos Clinic, Gandrup, North Denmark
  - Odense Universitetshospital, Odense
  - Sanos Clinic Vejle, Vejle
- France (3):
  - Hôpital Saint- Philibert, Lille
  - Hôpital Tenon, Paris
  - CHU Toulouse Rangueil, Toulouse
- United Kingdom (4):
  - Synexus Birmingham, Birmingham
  - North Bristol NHS Trust, Bristol
  - Addenbrookes, Cambridge
  - Synexus Merseyside, Liverpool

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 82 participants were enrolled, one was excluded to screening failure before randomization. Therefore, only 81 subjects are included in the groups.
Groups:
- Investigational Device First Then Comparator Device: Investigational device - newly developed intermittent catheter: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
  Comparator: The study protocol pre-specified that the comparator group would combine an equal split between two similar conventional-eyelet catheters, to achieve a comparator arm representing this class of devices as closely as possible. Subjects were randomized to receive either one of the comparator products; either SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked products produced by Coloplast.
  Comparator device #1 - SpeediCath Eve:
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use. Details on the comparator devices are as follows:
  Comparator device #2 - SpeediCath Compact Plus Female:
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
- Comparator Device First Then Investigational Device: Comparator: The study protocol pre-specified that the comparator group would combine an equal split between two similar conventional-eyelet catheters, to achieve a comparator arm representing this class of devices as closely as possible. Subjects were randomized to receive either one of the comparator products; either SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked products produced by Coloplast.
  Comparator device #1 - SpeediCath Eve:
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use. Details on the comparator devices are as follows:
  Comparator device #2 - SpeediCath Compact Plus Female:
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
  Investigational device - newly developed intermittent catheter: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
Period: First Intervention (14 Days)
Arm/Group | Investigational Device First Then Comparator Device | Comparator Device First Then Investigational Device
Started | 40 | 41
Comparator #1 | 20 | 20
Comparator #2 | 20 | 21
Completed | 39 | 40
Not Completed | 1 | 1
Period: Second Intervention (14 Days)
Arm/Group | Investigational Device First Then Comparator Device | Comparator Device First Then Investigational Device
Started | 39 | 40
Comparator #1 | 19 | 19
Comparator #2 | 20 | 21
Completed | 37 | 39
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population Baseline Measures: As this study was a crossover study, each participant underwent catheterizations with both the investigational device and the comparator device. The study consisted of three study visits (V1-V3) and two 2-week test periods at home (T1 and T2). Visit 1 included subject enrollment, and randomization. Randomization was done centralized, randomly assigning subjects to two intervention sequences. Hence, the first group used the investigational device during the first test period at home (T1) and at the first follow-up visit (V2). Subsequently, the comparator device was tested during the next test period at home (T2) followed by a visit 3 which also terminated the study. The second group tested the devices in reversed order. The total study duration was approximately 4 weeks for the individual subject
Arm/Group | Total ITT Population Baseline Measures
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 55
  United Kingdom | 14
  France | 12

OUTCOME MEASURES:

1. Primary Outcome: Residual Volume at 1st Flow-stop (Catheterisation Performed by HCP)
Description: Residual volume at 1st flow-stop i.e., post catheterisation volume minus volume at 1st flow-stop, both derived from a catheterisation profile (catheterisation performed by a healthcare professional)
Time Frame: Tested at site visit after 14 days of device home use.
Population: The study protocol pre-specified that the comparator arm of the study would combine an equal split between two similar conventional-eyelet catheters, to achieve a comparator arm representing this class of devices as closely as possible. Subjects were randomized to receive either one of the comparator products; either SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked products produced by Coloplast.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters
Groups:
- Investigational Device - Newly Developed Intermittent Catheter: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (CH12 and CH14) for urinary drainage. The investigational device is for single use.
  Randomization will decide the order of investigational device/comparator device and which of the two comparator devices the subject will receive in the comparator study period.
  Investigational device - newly developed intermittent catheter: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
- Comparator Device: The comparator device used was randomized evenly between SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked Coloplast products and both are conventional-eyelet compact female catheters. The similarity of these products were the reason for their combination into one group.
  Comparator device #1 - SpeediCath Eve: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
  Comparator device #2 - SpeediCath Compact Plus Female: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device
Number analyzed (Participants) | 79 | 79
milliliters | 23.22 [4.65 to 41.80] | 15.87 [6.09 to 25.65]

2. Secondary Outcome: Number of Flow-stops (Catheterisation Profile, Catheterisation Performed by HCP)
Description: Number of flow-stop episodes derived from a catheterisation profile (catheterisation performed by a healthcare professional)
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of flow-stops
Groups:
- Comparator Device (#1 OR #2): The comparator device used was randomized evenly between SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked Coloplast products and both are conventional-eyelet compact female catheters. The similarity of these products were the reason for their combination into one group.
  Comparator device #1 - SpeediCath Eve: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
  Comparator device #2 - SpeediCath Compact Plus Female: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 79 | 79
Number of flow-stops | 0.21 [0.10 to 0.44] | 0.57 [0.39 to 0.82]

3. Secondary Outcome: Number of Flow-stops (Catheterisation Profile, Self-catheterisation)
Description: Number of flow-stop episodes derived from a catheterisation profile (self-catheterisation)
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of flow-stops
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 79 | 79
Number of flow-stops | 0.28 [0.12 to 0.63] | 0.71 [0.52 to 0.95]

4. Secondary Outcome: Residual Volume at 1st Flow-stop
Description: Residual volume at 1st flow-stop i.e., post catheterisation volume minus volume at 1st flow-stop, both derived from a catheterisation profile (self-catheterisation)
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 79 | 79
milliliters | 19.88 [5.73 to 34.04] | 27.77 [12.14 to 43.40]

5. Secondary Outcome: Average Residual Volume Post Catheterisation (Bladder Scan)
Description: Average residual volume post catheterisation measured with the BladderScanner (triplicate measurements)
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: milliliters
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 79 | 79
milliliters
  HCP-led catheterisation | 4.8 (16.4) | 12.0 (40.4)
  Self-catheterisation | 7.7 (13.9) | 9.3 (20.5)

6. Secondary Outcome: Number of Adverse Events
Description: Number of Adverse events (number)
Time Frame: From Week 0-4
Population: as for outcome 1
Measure: Number; unit: Adverse events
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 81 | 81
Adverse events | 10 | 13

7. Other Pre Specified Outcome: Exploratory: Perception Questionnaire, Handling
Description: Perception questions evaluated on a 5-point scale assessed on V2 and V3 (perception questionnaire). Perception questionary based on perception of catheterisations in test period leading up to the visit
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 78 | 77
Participants
  1. How is it to use the catheter?: Difficult | 3 | 11
  1. How is it to use the catheter?: Easy | 17 | 21
  1. How is it to use the catheter?: Neither Difficult nor Easy | 1 | 7
  1. How is it to use the catheter?: Very difficult | 0 | 0
  1. How is it to use the catheter?: Very easy | 57 | 38
  1. How is it to use the catheter?: Don't know | 0 | 0
  2. How is it to open the catheter?: Difficult | 2 | 15
  2. How is it to open the catheter?: Easy | 23 | 26
  2. How is it to open the catheter?: Neither Difficult nor Easy | 7 | 8
  2. How is it to open the catheter?: Very difficult | 0 | 3
  2. How is it to open the catheter?: Very easy | 46 | 25
  2. How is it to open the catheter?: Don't know | 0 | 0
  3. How is it to insert the catheter?: Difficult | 2 | 7
  3. How is it to insert the catheter?: Easy | 18 | 29
  3. How is it to insert the catheter?: Neither Difficult nor Easy | 5 | 7
  3. How is it to insert the catheter?: Very difficult | 1 | 1
  3. How is it to insert the catheter?: Very easy | 52 | 33
  3. How is it to insert the catheter?: Don't know | 0 | 0
  4. How is it to empty the bladder?: Difficult | 3 | 2
  4. How is it to empty the bladder?: Easy | 19 | 35
  4. How is it to empty the bladder?: Neither Difficult nor Easy | 5 | 10
  4. How is it to empty the bladder?: Very difficult | 0 | 2
  4. How is it to empty the bladder?: Very easy | 51 | 28
  4. How is it to empty the bladder?: Don't know | 0 | 0
  5. How is it to handle the catheter during insertion?: Difficult | 3 | 8
  5. How is it to handle the catheter during insertion?: Easy | 24 | 22
  5. How is it to handle the catheter during insertion?: Neither Difficult nor Easy | 5 | 15
  5. How is it to handle the catheter during insertion?: Very difficult | 1 | 1
  5. How is it to handle the catheter during insertion?: Very easy | 45 | 31
  5. How is it to handle the catheter during insertion?: Don't know | 0 | 0
  6. How is it to re-close the catheter?: Difficult | 6 | 15
  6. How is it to re-close the catheter?: Easy | 34 | 16
  6. How is it to re-close the catheter?: Neither Difficult nor Easy | 6 | 9
  6. How is it to re-close the catheter?: Very difficult | 2 | 10
  6. How is it to re-close the catheter?: Very easy | 27 | 25
  6. How is it to re-close the catheter?: Don't know | 3 | 2

8. Other Pre Specified Outcome: Exploratory: Perception Questionnaire, Confidence, Sensation, Satisfaction
Description: as for outcome 7
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 78 | 77
Participants
  7. The catheter is discreet: Agree | 19 | 21
  7. The catheter is discreet: Disagree | 1 | 10
  7. The catheter is discreet: Don't know | 0 | 0
  7. The catheter is discreet: Neither disagree nor agree | 7 | 8
  7. The catheter is discreet: Not applicable (lack of sensation) | 0 | 0
  7. The catheter is discreet: Strongly agree | 50 | 34
  7. The catheter is discreet: Strongly disagree | 1 | 4
  8. The catheter is hygienic to use: Agree | 20 | 18
  8. The catheter is hygienic to use: Disagree | 2 | 9
  8. The catheter is hygienic to use: Don't know | 0 | 0
  8. The catheter is hygienic to use: Neither disagree nor agree | 2 | 9
  8. The catheter is hygienic to use: Not applicable (lack of sensation) | 0 | 0
  8. The catheter is hygienic to use: Strongly agree | 50 | 40
  8. The catheter is hygienic to use: Strongly disagree | 4 | 1
  9. It is fast to empty my bladder completely using this catheter: Agree | 22 | 30
  9. It is fast to empty my bladder completely using this catheter: Disagree | 5 | 6
  9. It is fast to empty my bladder completely using this catheter: Don't know | 0 | 1
  9. It is fast to empty my bladder completely using this catheter: Neither disagree nor agree | 15 | 18
  9. It is fast to empty my bladder completely using this catheter: Not applicable (lack of sensation) | 0 | 0
  9. It is fast to empty my bladder completely using this catheter: Strongly agree | 34 | 17
  9. It is fast to empty my bladder completely using this catheter: Strongly disagree | 2 | 5
  10. I feel the catheter has a sufficient length to empty my bladder completely: Agree | 16 | 35
  10. I feel the catheter has a sufficient length to empty my bladder completely: Disagree | 6 | 3
  10. I feel the catheter has a sufficient length to empty my bladder completely: Don't know | 1 | 0
  10. I feel the catheter has a sufficient length to empty my bladder completely: Neither disagree nor agree | 5 | 10
  10. I feel the catheter has a sufficient length to empty my bladder completely: Not applicable (lack of sensation) | 0 | 0
  10. I feel the catheter has a sufficient length to empty my bladder completely: Strongly agree | 48 | 27
  10. I feel the catheter has a sufficient length to empty my bladder completely: Strongly disagree | 2 | 2
  11. I feel confident the catheter empties my bladder completely: Agree | 24 | 29
  11. I feel confident the catheter empties my bladder completely: Disagree | 6 | 11
  11. I feel confident the catheter empties my bladder completely: Don't know | 1 | 0
  11. I feel confident the catheter empties my bladder completely: Neither disagree nor agree | 4 | 12
  11. I feel confident the catheter empties my bladder completely: Not applicable (lack of sensation) | 0 | 0
  11. I feel confident the catheter empties my bladder completely: Strongly agree | 43 | 22
  11. I feel confident the catheter empties my bladder completely: Strongly disagree | 0 | 3
  12. I don't worry about urine left in my bladder using this catheter: Agree | 15 | 30
  12. I don't worry about urine left in my bladder using this catheter: Disagree | 5 | 11
  12. I don't worry about urine left in my bladder using this catheter: Don't know | 0 | 0
  12. I don't worry about urine left in my bladder using this catheter: Neither disagree nor agree | 9 | 8
  12. I don't worry about urine left in my bladder using this catheter: Not applicable (lack of sensation) | 0 | 0
  12. I don't worry about urine left in my bladder using this catheter: Strongly agree | 47 | 24
  12. I don't worry about urine left in my bladder using this catheter: Strongly disagree | 2 | 4
  13. I feel confident using the catheter: Agree | 13 | 26
  13. I feel confident using the catheter: Disagree | 4 | 5
  13. I feel confident using the catheter: Don't know | 0 | 0
  13. I feel confident using the catheter: Neither disagree nor agree | 3 | 7
  13. I feel confident using the catheter: Not applicable (lack of sensation) | 0 | 0
  13. I feel confident using the catheter: Strongly agree | 57 | 35
  13. I feel confident using the catheter: Strongly disagree | 1 | 4
  14. It is gentle to insert the catheter: Agree | 19 | 32
  14. It is gentle to insert the catheter: Disagree | 2 | 5
  14. It is gentle to insert the catheter: Don't know | 0 | 0
  14. It is gentle to insert the catheter: Neither disagree nor agree | 1 | 3
  14. It is gentle to insert the catheter: Not applicable (lack of sensation) | 3 | 3
  14. It is gentle to insert the catheter: Strongly agree | 51 | 29
  14. It is gentle to insert the catheter: Strongly disagree | 2 | 5
  15. It is gentle to empty the bladder: Agree | 16 | 30
  15. It is gentle to empty the bladder: Disagree | 1 | 6
  15. It is gentle to empty the bladder: Don't know | 0 | 0
  15. It is gentle to empty the bladder: Neither disagree nor agree | 3 | 3
  15. It is gentle to empty the bladder: Not applicable (lack of sensation) | 3 | 2
  15. It is gentle to empty the bladder: Strongly agree | 55 | 32
  15. It is gentle to empty the bladder: Strongly disagree | 0 | 4
  16. It is gentle to withdraw the catheter: Agree | 18 | 28
  16. It is gentle to withdraw the catheter: Disagree | 3 | 7
  16. It is gentle to withdraw the catheter: Don't know | 0 | 0
  16. It is gentle to withdraw the catheter: Neither disagree nor agree | 1 | 5
  16. It is gentle to withdraw the catheter: Not applicable (lack of sensation) | 2 | 4
  16. It is gentle to withdraw the catheter: Strongly agree | 54 | 26
  16. It is gentle to withdraw the catheter: Strongly disagree | 0 | 7
  17. I feel pinching/stinging during catheterization using this catheter: Agree | 3 | 11
  17. I feel pinching/stinging during catheterization using this catheter: Disagree | 27 | 24
  17. I feel pinching/stinging during catheterization using this catheter: Don't know | 0 | 0
  17. I feel pinching/stinging during catheterization using this catheter: Neither disagree nor agree | 2 | 5
  17. I feel pinching/stinging during catheterization using this catheter: Not applicable (lack of sensation) | 3 | 4
  17. I feel pinching/stinging during catheterization using this catheter: Strongly agree | 1 | 7
  17. I feel pinching/stinging during catheterization using this catheter: Strongly disagree | 42 | 26
  18. I am satisfied with the catheter: Agree | 22 | 30
  18. I am satisfied with the catheter: Disagree | 7 | 13
  18. I am satisfied with the catheter: Don't know | 0 | 0
  18. I am satisfied with the catheter: Neither disagree nor agree | 6 | 9
  18. I am satisfied with the catheter: Not applicable (lack of sensation) | 0 | 0
  18. I am satisfied with the catheter: Strongly agree | 41 | 16
  18. I am satisfied with the catheter: Strongly disagree | 2 | 9
  19. I would like to use the catheter in the future: Agree | 15 | 22
  19. I would like to use the catheter in the future: Disagree | 10 | 12
  19. I would like to use the catheter in the future: Don't know | 1 | 1
  19. I would like to use the catheter in the future: Neither disagree nor agree | 8 | 13
  19. I would like to use the catheter in the future: Not applicable (lack of sensation) | 0 | 0
  19. I would like to use the catheter in the future: Strongly agree | 39 | 11
  19. I would like to use the catheter in the future: Strongly disagree | 5 | 18
  20. I would recommend the catheter to others: Agree | 16 | 24
  20. I would recommend the catheter to others: Disagree | 3 | 11
  20. I would recommend the catheter to others: Don't know | 3 | 1
  20. I would recommend the catheter to others: Neither disagree nor agree | 13 | 16
  20. I would recommend the catheter to others: Not applicable (lack of sensation) | 0 | 0
  20. I would recommend the catheter to others: Strongly agree | 41 | 12
  20. I would recommend the catheter to others: Strongly disagree | 2 | 13

9. Post Hoc Outcome: Response to Treatment, Residual Volume of Urine at First Flow-stop Under 10 Milliliter
Description: Responder analysis involved testing the proportion of all catheterisations which achieved a residual volume of urine at first flow-stop of less than 10 milliliter
  In this clinical investigation, responder analyses were introduced as an expansion of the data analyses due to the few extreme RV1 values, which presented a challenge to the predetermined statistical model. (see 'limitations and caveats' section for further details). Responder analyses evaluated the proportion of patients who achieved the positive treatment response threshold, highlighting individual patient responses rather than average effects across the entire population. Successful treatment responses were defined as individuals who achieved the desired outcome of catheterisation, i.e., complete and effective bladder emptying without repositioning, in terms flow-stops defined as zero flow-stops and in terms of complete emptying of the bladder was defined as an RV1<10 mL.
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of catheterisations
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 79 | 79
percentage of catheterisations | 83 [76 to 89] | 71 [63 to 78]

10. Post Hoc Outcome: Response to Treatment, 0 Flow-stops
Description: Responder analysis involved testing the proportion of all catheterisations which did not experience any flow-stops.
  In this clinical investigation, responder analyses were introduced as an expansion of the data analyses due to the few extreme RV1 values, which presented a challenge to the predetermined statistical model. (see 'limitations and caveats' section for further details). Responder analyses evaluated the proportion of patients who achieved the positive treatment response threshold, highlighting individual patient responses rather than average effects across the entire population. Successful treatment responses were defined as individuals who achieved the desired outcome of catheterisation, i.e., complete and effective bladder emptying without repositioning, in terms flow-stops defined as zero flow-stops and in terms of complete emptying of the bladder was defined as an RV1<10 mL.
Time Frame: Tested at site visit after 14 days of device home use.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of catheterisations
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device (#1 OR #2)
Number analyzed (Participants) | 79 | 79
percentage of catheterisations | 87 [80 to 92] | 57 [48 to 65]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: The study protocol pre-specified that the comparator arm of the study would combine an equal split between two similar conventional-eyelet catheters, to achieve a comparator arm representing this class of devices as closely as possible. Subjects were randomized to receive either of the comparator products; either SpeediCath Eve or SpeediCath Compact Plus Female. This specification also extended to the collection of adverse events, reporting adverse events of the comparator in combination.
Groups:
- Comparator Device: The study protocol pre-specified that the comparator arm of the study would combine an equal split between two similar conventional-eyelet catheters, to achieve a comparator arm representing this class of devices as closely as possible. Subjects were randomized to receive either one of the comparator products; either SpeediCath Eve or SpeediCath Compact Plus Female (CH12 and CH14). Both comparators are CE marked products produced by Coloplast.
  Comparator device #1 - SpeediCath Eve:
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use. Details on the comparator devices are as follows:
  Comparator device #2 - SpeediCath Compact Plus Female:
  Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The comparator device is for single use.
Arm/Group | Investigational Device - Newly Developed Intermittent Catheter | Comparator Device
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 10/81 | 13/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Device - Newly Developed Intermittent Catheter (N=81) | Comparator Device (N=81)
Urinary tract infection (Renal and urinary disorders) | 3 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Tingling sensation when urinating (Renal and urinary disorders) | 0 | 1
Urinary discomfort (Renal and urinary disorders) | 0 | 1
Common cold (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Muscle pain in back (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle pain in left leg (Musculoskeletal and connective tissue disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 2
Tooth ache (General disorders) | 1 | 0
Fall (General disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Flank pain (General disorders) | 0 | 1
Vasovagal syncope (Vascular disorders) | 0 | 1
Foul smelling urine (Renal and urinary disorders) | 0 | 1
Herpes labial (Infections and infestations) | 0 | 1
Pyelonefritis (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The natural distribution of residual volume at 1st flow-stop values skews positively. This carries a high risk of influence by random occurrences of extreme values. These can occur without systematic relation to product or subject and can obscure interpretability of the analysis. To counter this effect, post hoc responder analyses were included, testing the benefit of treatment through the proportion of individuals who achieve the desired outcome, i.e., complete and effective bladder drainage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT05814211/Prot_SAP_000.pdf